CLINICAL TRIAL: NCT03884907
Title: Multicentric Observational Study on the Use of a Human Bone Graft in Austin Procedure of Hallux Valgus Correction
Brief Title: Human Bone Graft for Hallux Valgus Correction According to the Austin Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Wels-Grieskirchen (Other)
Collaborators: Surgebright Gmbh (Industry)
Responsible Party: Principal Investigator, Dr. Thorsten Huber, Assistent surgeon, team member of the foot team, Klinikum Wels-Grieskirchen
Other Study IDs: 1032/2018
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Hallux Valgus
Keywords: human bone graft screw; foot and ankle surgery; hallux valgus deformity
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: The patients will receive human bone graft screws surgically — All patients undergo Hallux valgus correction according to the Austin procedure using human bone graft screws.

SUMMARY:
This observational study is to document the application of a human bone graft in the surgical repair of hallux valgus deformity and its subsequent healing process.

DETAILED DESCRIPTION:
For the treatment of bone fractures metal screws have been used for decades. Removal of material is the major disadvantage of conventional osteosynthesis and requires a second intervention, with all the complications and risks for each patient. Moreover, the metal screw disturbs as foreign material in the bone and irritates the surrounding soft tissue.

In order to overcome the drawbacks of metal screws human bone screw grafts can be used instead representing a biodegradable osteosynthesis material with ideal material properties.

The bone graft helps to create a solid, bony connection. This connection leads to an extension, a bone remodeling, bone installation and optimal reparation process in the affected area.

This observational study is being conducted in order to overcome the lack of systematic research to objectively confirm the benefits of the product.

In total 50 patients will be enrolled in this study in several centers in Austria This observational study will use Shark Screw® grafts manufactured by two tissue banks, the Austrian Tissue Bank surgebright and the German Institute for Cell and Tissue Replacement (DZIG). The Shark Screw® grafts were approved by the competent Austrian authority (AGES) in 2016.

All patients participating in this observational study, due to a medical indication, undergo Hallux valgus correction according to the Austin procedure using the bone screws mentioned above.

A 12 month postoperative observation period is set. Five routine follow-up examinations including clinical examination and x-ray analysis will be performed. In case the an additional routine follow-up examination is necessary for clinical reason within 24 month post-operative, the patient remains in the study.

ELIGIBILITY:
Inclusion Criteria:

* Indication for the use of a human bone graft in the surgical treatment of Hallux valgus treatment using Austin procedure
* legal capability of adults
* Written consent to participation in the study after previous written and oral education
* Age ≥ 18 years

Exclusion Criteria:

* Insufficient knowledge of the German language
* Alcohol and drug abuse
* Pregnant or breastfeeding woman
* Foreseeable compliance issues
* Neoplastic diseases, malignant bone tumors, rheumatoid arthritis
* Active osteomyelitis
* Ulcerations in the area of the skin of the surgical area
* Revision surgery after primary Hallux valgus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from all participating sites scheduled for a Hallux valgus correction using the Austin procedure with human bone graft screws get information about this observational study and have the possibility to participate.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-08-21 (Estimated); Study Completion 2020-03-21 (Estimated)

PRIMARY OUTCOMES:
incidence of surgical revisions | 1 year
  Was a surgical revision done postoperatively? YES/NO
incidence of loosening of the screw | 1 year
  based on x-rays: Is a loosening of the screw visible? YES/NO
incidence of cracking of the screw | 1 year
  based on x-rays: Is a cracking of the screw visible? YES/NO
Hallux valgus angle | 1 year
  based on x-rays: What ist he Hallux valgus angle? °
Intermetatarsal angle | 1 year
  based on x-rays: What is the intermetatarsal angle? °
incidence of postoperative pseudoarthrosis | 1 year
  based on x-rays or MRI: Is a postoperative pseudoarthrosis visible? YES/NO
evaluation postoperative pain (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = no pain - 100mm = worst imaginable pain). A higher score indicates more pain.
duration of postoperative job-related incapacity | 1 year
  evaluation of duration

SECONDARY OUTCOMES:
Patient satisfaction (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = very satisfied - 100mm = not satisfied at all). A higher score indicates less satisfaction.
Assessment according to the AOFAS score | 1 year
  AOFAS (American Orthopaedic Foot and Ankle Society) Score evaluates the functional impairments of food and ankle. The AOFAS score consists of 8 questions in the categories pain (40 points), function (6 questions, total 45 points) and alignment (15 points). The scores of all questions are summed up to the total score. The maximum score is 100, where 100 is the best outcome and 0 is the worst outcome. All questions are to be answered relating to the previous week.

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - A.ö. Bezirkskrankenhaus St. Johann in Tirol, Sankt Johann in Tirol, Tyrol
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria

IPD SHARING:
Plan to Share IPD: Undecided